CLINICAL TRIAL: NCT02985619
Title: Randomized Trial Evaluating Bevacizumabe or Triamcinolone for Persistent Diabetic Macular Edema
Brief Title: Bevacizumabe or Triamcinolone for Persistent Diabetic Macular Edema
Acronym: BEVATAAC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Murilo Wendeborn Rodrigues Junior, USP Ribeirao Preto, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.599.864
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IVB randomised group I (Active Comparator): Randomised patients [intravitreal bevacizumab (IVB) group I] with central foveal thickness >300µm on OCT will be submitted to 6 months treatment with 0.05ml (1.25mg) intravitreous injection of Bevacizumabe "prn" (pro re nata, or as needed), with monthly visits for central subfoveal thickness map more than 300µm by Optic Coherence Tomography. Care will be take in all cases to insure that the needle do not touch the lids or lashes. Bevacizumab (1.25 mg/0.05 cc; F. Hoffmann- La Roche Ltd., Basel, Switzerland) will be inject into the vitreous cavity using a 29-gauge 0.5- inch needle insert through the superotemporal pars plana 3.0-3.5 mm posterior to the limbus.
  Interventions: Drug: Bevacizumab Injection [Avastin] (IVB-I)
- IVT randomised group II (Active Comparator): Randomised patients [intravitreal triamcinolone (IVT) group II] with central foveal thickness >300µm on OCT will be submitted to 6 months treatment with 0.03ml (1.20mg) intravitreous injection of triamcinolone each 3 months (prn, as needed) for central sufoveal thickness map more than 300µm by Optic Coherence Tomography. Care will be take in all cases to insure that the needle do not touch the lids or lashes. Triamcinolone (1.20 mg/ 0.03 cc; Opthaac, Ophthalmos, São Paulo, Brazil) will be inject into the vitreous cavity using a 29-gauge 0.5- inch needle insert through the superotemporal pars plana 3.0-3.5 mm posterior to the limbus.
  Interventions: Drug: Triamcinolone Acetonide 10mg/mL (IVT-II)
- IVB group III (not randomised) (Active Comparator): Patients with central foveal thickness ≤300µm at week visit 24 will be allocated to group III (IVB, intravitreal bevacizumab). So, it won't get IVB injection at week visit 24 due OCT regular thickness (≤300µm) but will do regular monthly follow-up visits and prn-IVB therapy if central foveal thickness >300µm on OCT until last visit of study (48 week-visit). Care will be take in all cases to insure that the needle do not touch the lids or lashes. Bevacizumab (1.25 mg/0.05 cc; F. Hoffmann- La Roche Ltd., Basel, Switzerland) will be inject into the vitreous cavity using a 29-gauge 0.5- inch needle insert through the superotemporal pars plana 3.0-3.5 mm posterior to the limbus.
  Interventions: Drug: Bevacizumab Injection [Avastin] (IVB-III)

INTERVENTIONS:
Drug: Bevacizumab Injection [Avastin] (IVB-I) — 0,05ml intravitreal injection
  Other Names: Avastin®
  Arms: IVB randomised group I
Drug: Triamcinolone Acetonide 10mg/mL (IVT-II) — 0,03ml intravitreal injection
  Other Names: OPTHTAAC®
  Arms: IVT randomised group II
Drug: Bevacizumab Injection [Avastin] (IVB-III) — 0,05ml intravitreal injection
  Other Names: Avastin®
  Arms: IVB group III (not randomised)

SUMMARY:
Background: Diabetic macular edema (DME) shows a sustained functional and morphologic response to anti-vascular endothelial growth factor (VEGF) drugs, but the optimal approach for persistent macular edema still in debate.

Purpose: To evaluate 24-week visual and anatomical effects of intravitreal bevacizumabe or triamcinolone in patients who have residual edema after 24-weeks to "pro re nata"(prn) intravitreal bevacizumabe therapy.

Methods: This study will enroll a total of 100 DME eyes. Each patient will receive "prn" bevacizumabe therapy throughout 24 weeks. At week 24, patients who have recurrent or persistent edema were randomized 1:1 to Group 1 (prn bevacizumane) or Group 2 (prn triamcinolone). Patients with no recurrent or persistent edema at week 24 will comprise to Group 3 and continue receive prn bevacizumabe. Prn treatment was administered when central subfield thickness of the macula (CST) > 300 µm and/or there are intraretinal cystoid spaces in the fovea. Study visits will occur every 4 weeks with the endpoint at week 48. At each visit, patients will have an eye exam and CST, best-corrected visual acuity (BCVA), and intraocular pressure (IOP) were assessed. Fundus photography and fluorescein angiography will also perform at baseline, week 16, week 40, and week 48. All patients will resume standard care after exiting.

DETAILED DESCRIPTION:
Methods Study Design. The current study is a prospective randomized clinical trial registered at ClinicalTrials.gov (NCT02985619). The study protocol adhered to the tenets of the Declaration of Helsinki and was approved by the local Institutional Review Board, research ethics committee of School of Medicine of Ribeirão Preto at University of Sao Paulo. All patients will give inform consent signature before entering one year study and will evaluate in the Retina Section of Department of Ophthalmology, School of Medicine of Ribeirao Preto of the University of Sao Paulo with center-involved DME in at least 1 eye. Recruiting phase will be consider the first 6 months. All patients with diagnostic of DME in at least 1 eye from July 2016 to December 2016 will invite to participate in the study.

Study Population. Inclusion criteria. Inclusion criteria are as follows: (1) Eligible participants are age 18 years old with diabetes mellitus (type 1 or 2); (2) center-involved DME, defined as a central subfield thickness >300 µm on spectral domain optical coherence tomography (SD-OCT), despite of macular laser photocoagulation, cataract surgery and intraocular injection performed at least 4 months previously; (3) best-corrected ETDRS visual acuity (BCVA) measurement between 0.3 logMAR (Snellen equivalent: 20/32) and 1.3 logMAR (Snellen equivalent: 20/400); (4) signed informed consent. Exclusion criteria. Exclusion criteria were: (1) vitreo-macular traction on SD-OCT; (2) proliferative diabetic retinopathy needing panretinal photocoagulation (PRP) or anticipated to need PRP in the next 12 months; (3) macular capillary dropout on fluorescein angiography; (4) history of glaucoma or ocular hypertension (defined as an intraocular pressure higher than 25 mm Hg); (5) an ocular condition (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (eg, retinal vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc); (6) systemic corticosteroid therapy; (7) any condition that, in the opinion of the investigator, might preclude follow-up throughout the study period; (8) Recent (within 3 months) thromboembolic events including acute myocardial infarction (MI) and cerebrovascular accident (CVA); (9) Other Clinical trial participation in the last 30 days.

Randomization and Intervention. After eligibility phase, subjects with center-involving DME will enroll and undergo comprehensive ophthalmologic evaluation at baseline and every 4 weeks up to week 48. Patients will receive monthly prn 1.25 mg (0.05 cc) IVB throughout 24 weeks if central subfield thickness (CSFT) will great than 300 µm. At week 24, patients who has recurrent or persistent edema (CSFT>300) will randomize 1:1 to Group 1 (prn IVB therapy) or Group 2 (quarterly IVT therapy). Randomization will be do from binomial distribution with parameters that it enters as function arguments. Patients with no recurrent or persistent edema (CSFT≤300µm) at 24-week will comprise to Group 3 and continue receiving prn IVB therapy. If patient have edema in both eyes and the patient agree to treat both eyes, 1 eye will receive the random treatment according to a computer-generate sequence and the contralateral eye will receive the other therapy option on the next day; thus if an eye was randomized to the IVB group I, the contralateral eye will allocate to the IVT group II and the reverse will also true.

Examination Procedures and follow-up. Each patient will receive a detailed ophthalmologic examination including measurement of BCVA according to the standardized ETDRS refraction protocol using a retroilluminate Lighthouse for the Blind distance visual acuity test chart (using modified ETDRS charts 1, 2, and R; Precision Vision, IL), as well as applanation tonometry, slit-lamp biomicroscopic examination, indirect fundus examination, and fluorescein angiography using high-resolution angiography (HRA; Heidelberg Engineering, Heidelberg, Germany). SD-OCT evaluation (HRA-OCT; Heidelberg Engineering) will be performe in all patients, and retinal thickness measurements will be acquire using a standard 20, 15-degree raster scan protocol. CSFT values will be calculate automatically as the average thickness of a central macular region 1000 mm in diameter centered on the patient's foveola by built-in Heidelberg software using retinal map analysis. Patients will schedule for follow-up examinations at monthly intervals. At these visits the BCVA will be determined after ETDRS refraction and complete ophthalmic examination similar to baseline valuations with the exception of fluorescein angiography schedule at baseline and week 36.

Antiglaucomatous eyedrops criteria. Intraocular pressure (IOP) ≥ 25 mmHg and/or 10mmHg increased from baseline measurement will be adopt to initiate anti-glaucomatous eyedrops.

Intravitreal Injection. All injections will be were performed using topical proparacaine drops under sterile conditions (eyelid speculum and povidone-iodine). Topical antibiotics will not use before the day of injection. Before the injection are perform, the eyelids will scrubb with 10% povidone-iodine, and 5% povidone-iodine drops will be apply to the conjunctiva. The time between application of 5% povidone-iodine solution to the conjunctiva and administration of the intravitreal injection will be 2 minutes. Povidone-iodine will be was apply to the conjunctiva directly over the intended injection site. Care will be take in all cases to insure that the needle do not touch the lids or lashes. Bevacizumab (1.25 mg/0.05 cc; F. Hoffmann- La Roche Ltd., Basel, Switzerland) or Triamcinolone (1.20 mg/ 0.03 cc; Opthaac, Ophthalmos, São Paulo, Brazil) will be inject into the vitreous cavity using a 29-gauge 0.5- inch needle insert through the superotemporal pars plana 3.0-3.5 mm posterior to the limbus.25 After the injection, central retinal artery perfusion will be confirm with indirect ophthalmoscopy. Patients will instruct to instill 1 drop of 0.3% ciprofloxacin into the inject eye 4 times daily for 1 week after the procedure.

Retreatment Protocol. Retreatment with the originally assign treatment is perform monthly if central subfield thickness is great than 300 µm.

Rescue Therapy. Before randomization, all patients will receive prn-IVB and if, after 3 consecutive visits, there will be not a reduction in CST of at least 10% or an increase in BCVA of at least 5 ETDRS letters score when compare with baseline, the patient can continue with the same intravitreal medication for an additional 3 consecutive visits or discontinue treatment. After randomization, a similar strategy is used as rescue therapy for all 3 groups.

Outcomes. Primary outcome measure: Mean change in CSFT from baseline to week 48. Secondary outcomes measures: Mean change in BCVA from baseline to week 48; mean change in IOP at any visit; lens status changes, mean number of intravitreous injections Sample Size. Sample size and powering is base on a previous clinical trial on bevacizumab use for diabetic macular edema, where a mean change observed in central subfield thickness from baseline was 130 mm with a standard deviation of 122 μm. Therefore, to have 80% power to detect a difference of 50 μm between central subfield thickness change found in both groups, the sample size require in each group was 25 eyes. Thirty eyes per treatment group is require if one assume a 10% dropout rate. With this sample size, there is a 20% chance for a failure to detect a true mean difference of at least 50 μm between the treatment groups (type I error), or for an incorrect conclusion that a difference of at least 50 μm exists between the treatment groups (type II error).

Statistical Analysis. BCVA and central subfield thickness measured at each follow-up visit will be compare with baseline BCVA and CSFT values for within- and between-group comparisons, which is perform using multiple analysis of variance (MANOVA) for repeated measurements. Proportions of eyes with central subfield thickness ≤ 300 mm is compare using the likelihood ratio x2 test. In addition, a multivariate analysis comparing BCVA and CSFT outcomes in the prn-IVB group and qIVT group is perform, considering number of injections, baseline BCVA, and CSFT as effects. A statistically significant effect is define if P < .05, and a trend towards significance is report if P < .1. Statistical analyses are performe using JMP 10.0.0 (2010; SAS Institute Inc, Cary, North Carolina, USA) software.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema with >300µm on central subfield macular thickness by OCT;
* Best corrected vision acuity minimum: 20/32 to 20/320;

Exclusion Criteria:

* Vitreomacular traction;
* Macular ischemia;
* Laser or injection therapy before 3 months to assign the protocol.\
* Pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
OCT measurements | 6 months.
  Optical Coherence Tomography measurements in the central subfield thickness between baseline and 6 months 1st endpoint.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-05-29): https://cdn.clinicaltrials.gov/large-docs/19/NCT02985619/Prot_SAP_ICF_000.pdf